CLINICAL TRIAL: NCT07406802
Title: Association Between Racket Stiffness and Lateral Epicondylalgia in Tennis Players: A Multicenter Observational Study
Brief Title: Association Between Racket Stiffness and Lateral Epicondylalgia in Tennis Players
Status: Not yet recruiting | Type: Observational
Sponsor: University of Oviedo (Other)
Responsible Party: Principal Investigator, Ruben Cuesta Barriuso, Principal Investigator, University of Oviedo
Other Study IDs: TENrig
Record Dates: First submitted 2026-02-05; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Tennis Elbow
Keywords: Tennis Elbow; Sports Injuries; Equipment Design; Pain Measurement
MeSH Terms: conditions — Tennis Elbow; Athletic Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observacional group: Adult tennis players in whom the association between racket stiffness and the presence of lateral epicondylalgia will be evaluated, including an analysis of the potential effect modification by sex and competitive level on this association.
  Interventions: Other: Adult tennis players

INTERVENTIONS:
Other: Adult tennis players — Adult tennis players in whom the association between racket stiffness and the presence of lateral epicondylalgia will be evaluated, including an analysis of the potential effect modification by sex and competitive level on this association.

SUMMARY:
Background. Lateral epicondylalgia is common in tennis and is associated with pain and functional limitation. Although racket stiffness has been experimentally linked to vibration transmission, its clinical association with this condition in tennis players remains insufficiently studied.

Objective. To evaluate the association between racket stiffness and the presence of lateral epicondylalgia in adult tennis players, and to examine the potential effect modification by sex and competitive level on this association.

Methods. An analytical observational study with a cross-sectional design will be conducted. A total of 200 athletes will be recruited. The primary outcome will be the presence of lateral epicondylalgia within the previous 12 months. Functional severity will be assessed using the Patient-Rated Tennis Elbow Evaluation Questionnaire. The main independent variable will be racket stiffness (RA/stiffness). Secondary variables will include string age, use of a vibration dampener, and exposure related to playing load and technique. Potential confounders will include sex, competitive level, age, anthropometric characteristics, smoking status, prior history of elbow pain, occupational ergonomics involving repetitive gripping (ISO 11228-3 criteria), sleep quality (Pittsburgh Sleep Quality Index), and racket characteristics. The prevalence of lateral epicondylalgia will be estimated, and multivariable logistic regression models will be used to assess the association between racket stiffness and lateral epicondylalgia, including interaction terms to evaluate effect modification by sex and competitive level.

Expected results. To determine the prevalence of lateral epicondylalgia in adult tennis players and to identify the association between racket stiffness and the presence of this condition, as well as the potential modifying effects of sex and competitive level.

ELIGIBILITY:
Inclusion Criteria:

* Tennis players aged 16 years or older.
* Regular tennis practice over the previous 12 months, defined as at least one weekly training or competition session.
* Habitual use of an adult tennis racket weighing more than 280 grams for training and competition for a minimum period of three months prior to data collection.
* Provision of written informed consent. Players with a history of elbow pain related to tennis practice will be eligible for inclusion and this information will be recorded as an independent clinical variable.

Exclusion Criteria:

* Players with a history of upper-limb surgery within the previous year.
* Athletes with a prior medical diagnosis of neurological or rheumatological disease that could affect the upper limb.
* Athletes who sustained an acute traumatic injury to the shoulder, elbow, or wrist within the six months preceding the study.
* Participants who fail to complete the study questionnaires correctly.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Adult tennis players
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2026-02-13 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-05-11 (Estimated)

PRIMARY OUTCOMES:
Measurement of Clinical of lateral epicondylalgia within the previous 12 months. | Screening visit
  Lateral epicondylalgia will be assessed using the Patient-Rated Tennis Elbow Evaluation (PRTEE) Questionnaire. This instrument evaluates pain and functional disability in individuals with lateral epicondylalgia. The questionnaire consists of 15 items. The total PRTEE score is transformed to a 0-100 scale, where 0 indicates no pain or disability and 100 represents the worst possible pain and functional impairment.

SECONDARY OUTCOMES:
Measurement of racket stiffness. | Screening visit
  Racket stiffness will be assessed using the measured stiffness value (RA) or stiffness index. As not all racket models report this parameter, when participants are unaware of the RA value, it will be determined based on the exact brand, model, and year of manufacture, and subsequently obtained from manufacturer catalogs or technical reference tables. The unit of measurement will be the RA rating (Racquet Analysis rating), also referred to as the stiffness index.
Measurement of string age. | Screening visit
  String age will be measured as the number of months since the last restringing. This variable will be used as a mechanical proxy for string condition, as commonly applied in biomechanical studies and technical-sport performance recommendations.
Measurement of vibration dampener use | Screening visit
  Vibration dampener use will be recorded as a dichotomous variable (yes/no). When applicable, the specific dampener model will be documented. This variable is a recognized modifier of the vibratory spectrum, as described in experimental studies.
Measurement of load exposure and playing technique | Screening visit
  In this variable, data will be collected on the number of weekly training hours (measured in hours/week).
Measurement of load exposure and technique. | Screening visit
  In this variable, data will be collected on the years of tennis practice (number of years).
Measurement of load exposure and technique. | Screening visit
  In this variable, data will be collected on the number of weekly matches (matches/week).
Measurement of load exposure and technique. | Screening visit
  In this variable, data will be collected on upper-limb dominance (right / left).
Measurement of load exposure and technique. | Screening visit
  In this variable, data will be collected on whether the athlete performs specific weekly upper-limb strength training (yes / no).
Measurement of load exposure and technique. | Screening visit
  In this variable, data will be collected on the number of weekly strength training hours.
Measurement of load exposure and technique. | Screening visit
  In this variable, data will be collected on backhand execution (one-handed / two-handed).
Measurement of load exposure and technique. | Screening visit
  In this variable, data will be collected on competitive level (occasional recreational (≤1 session/week; no tournaments); regular recreational (2-3 sessions/week; occasional local leagues); regional competitive

OTHER OUTCOMES:
Measurement of gender | Screening visit
  This will be the variable acting as an a priori effect modifier, with an RA×sex interaction term included in the models, given that sex-related differences in injury patterns have been reported in padel and contextual differences have
Measurement of competitive level | Screening visit
  This will be assessed using a dichotomous variable (Federated / Non-federated). This variable will act as a potential effect modifier (RA×competitive level), as exposure level, technique, and equipment differ between rec
Measurement of age | Screening visit
  Age will be measured in years
Measurement of body weight. | Screening visit
  This variable will be measured in kilograms (kg)
Measurement of height | Screening visit
  This variable will be measured in meters (m)
Measurement of smoking status | Screening visit
  Smoking status will be recorded as a dichotomous variable (yes/no). This variable is included because some studies have shown that individuals with a history of smoking present higher odds of developing the condition compared with controls.
Measurement of previous history of elbow pain | Screening visit
  This variable will be assessed using ISO 11228-3 screening criteria and temporal exposure. Three dichotomous items anchored to the ISO 11228-3 criteria for repetitive upper-limb tasks will be used, along with a quantification of exposure time in hours per week.
Measurement of sleep quality | Screening visit
  Sleep quality will be assessed using the Pittsburgh Sleep Quality Index. This scale measures global sleep quality over the previous month, including aspects such as sleep latency, duration, efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction. It consists of 19 items grouped into seven domains, with a total score ranging from 0 to 21 (higher scores indicate poorer sleep quality; scores >5 indicate poor sleep quality).

CONTACTS AND LOCATIONS:
Overall Officials: Rubén Cuesta-Barriuso, PhD, Principal Investigator — Universidad de Oviedo
Locations (1):
- Universidad de Oviedo, Oviedo, Principality of Asturias, Spain

IPD SHARING:
Plan to Share IPD: Undecided